CLINICAL TRIAL: NCT00078481
Title: Phase 1B Clinical Trial to Establish the Safety and Tolerability of a Multiple-Dose Regimen of Idebenone Administered to Patients With Friedreich's Ataxia
Brief Title: Phase 1 Trial of Idebenone to Treat Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040129; 04-N-0129
Record Dates: First submitted 2004-02-27; First posted 2004-03-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-04

CONDITIONS: Friedreich Ataxia
Keywords: Neurodegeneration; Anti-Oxidant; Neuropathy; Hereditary; Spinocerebellar; Friedreich Ataxia; FRDA
MeSH Terms: conditions — Friedreich Ataxia; Nerve Degeneration | interventions — idebenone

INTERVENTIONS:
Drug: Idebenone

SUMMARY:
This study will determine the highest amount of idebenone that can be taken without harmful side effects in children, teenagers, and adults with Friedreich's ataxia, a progressive degenerative disease that affects several body systems. Studies in France and Canada showed that patients with Friedreich's ataxia who took idebenone had a decrease in the size of their left ventricle (main pumping chamber of the heart), which is often enlarged in this disease. It is possible that idebenone may also prevent the progression of nervous system degeneration in Friedreich's ataxia.

Patients 5 years of age and older with Friedreich's ataxia may be eligible for this study. Candidates are screened with a blood test and review of their medical records, including genetic studies.

Participants undergo the following procedures during a 6-day hospital admission to the NIH Clinical Center:

* Placement of an intravenous catheter (plastic tube inserted into a vein) for collecting blood samples after drug administration
* Blood and urine tests
* Heart examination, including electrocardiogram (EKG), to assess heart function and size.
* Idebenone therapy: Patients take three tablets a day (at 7 AM, 1 PM and 7 PM) on days 2, 3 and 4 of hospitalization. Blood samples are collected through the IV tube at 0.5, 1, 2, 4, and 6 hours after the first dose on day 2, then at 1 hour after the first and third doses every day, and then at 1, 2, 4, 8, 12, 24, 36, and 48 hours after the last dose on day 4 to determine how the body uses and eliminates the drug.
* Monitoring for drug side effects: Patients have frequent checks of vital signs (blood pressure, pulse, temperature, breathing rate) and a brief physical examination to check for drug side effects from the start of drug therapy on day 2 until at least 43 hours after the last dose on day 4.

Patients who experience no difficulties are discharged from the hospital after the sixth day with a 1-month supply of medication to take 3 times a day at home. They are contacted by phone every 2 weeks while taking the medication to check side effects. Blood tests are also done every 2 weeks to check for any abnormalities.

DETAILED DESCRIPTION:
Background: Friedreich's ataxia (FRDA) is a progressive, autosomal recessive, multisystem degenerative disease for which there is currently no effective treatment. Recent studies have demonstrated that lipid-soluble antioxidants lead to a modest reversal of cardiomyopathy in patients with FRDA. It is possible that antioxidants may also prevent the progression of neurodegeneration.

Objective: This will be a phase 1B, unblinded trial examining the toxicity and tolerability of the antioxidant idebenone given as a multiple-dose regimen for a short inpatient course and then long term to patients with FRDA.

Study Population: We aim to enroll 15 patients divided evenly among three age cohorts: children (ages 5-11), adolescents (ages 12-17), and adults (age greater than or equal to 18).

Design: Our primary objective is to examine the tolerability of idebenone given at a dose of 60 mg/kg/day for 72 hours (total of 9 doses) in an inpatient setting (NIH Clinical Center). This dose is below the maximum dose examined (75 mg/kg/day) that was well tolerated with no dose-limiting toxicity (DLT) in our phase 1A (protocol# 01-N-0167) study. The 72 hour course represents 5.5 half-lives of the drug based upon previous studies of the drug in healthy human subjects and our phase 1A data, thereby allowing the serum concentration of the drug to reach steady-state levels. This multiple dose regimen will allow us to examine accumulation of the drug and to examine tolerability of the drug at a steady-state concentration. The patients will then be followed by inpatient monitoring for an additional 43 hours, representing 3.3 half-lives, to allow relatively complete elimination of the drug. If no adverse events are noted during the inpatient phase of the trial, patients will resume taking the drug on an outpatient basis for 1 month to determine long-term tolerability and compliance. Outpatients will be followed through phone interviews by the NIH research team along with routine blood work every 2 weeks. Our secondary objective is to document the pharmacokinetics, specifically the apparent distribution volume (Vd), elimination half-life (t1/2), elimination clearance (CLE), and steady-state concentrations (CSS) of idebenone during the inpatient phase of the study.

Outcome Parameters: Outcomes in this phase I trial are types and frequency of adverse events, if any, and compliance with the dosing regimen. Our secondary endpoint is pharmacokinetics of this dosing regimen.

Future Directions: We hope to follow these phase I studies with a multicenter, double-blinded, placebo-controlled phase III trial using an ataxia scale developed for FRDA as the primary endpoint.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of FRDA with confirmed FRDA mutations.

Age greater than or equal to five years.

No exposure to idebenone or coenzyme Q(10) for a period of at least one week before onset of the medication phase of the study.

Written, informed consent (and assent, if applicable).

EXCLUSION CRITERIA:

History of hypersensitivity reaction to idebenone or coenzyme Q(10).

Pregnant or lactating women. All women of child-bearing potential must have negative serum pregnancy prior to the medication phase of the study. If a minor has a positive pregnancy test, we will inform her but not inform her parents unless we are asked to by the minor.

Lactose intolerant individuals (because of the lactose content in the tablet ingredients).

Age less than five years old.

Platelet count, lymphocyte count or hemoglobin below the lower limit of normal.

Alkaline phosphatase, SGOT, or SGPT greater than 1.5 x the upper limit of normal. Bilirubin greater than 1.2 g/dl.

Creatinine greater than 1.5 x the upper limit of normal.

Clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2004-02; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Artuch R, Aracil A, Mas A, Colome C, Rissech M, Monros E, Pineda M. Friedreich's ataxia: idebenone treatment in early stage patients. Neuropediatrics. 2002 Aug;33(4):190-3. doi: 10.1055/s-2002-34494. PMID 12368988
- [Background] Babcock M, de Silva D, Oaks R, Davis-Kaplan S, Jiralerspong S, Montermini L, Pandolfo M, Kaplan J. Regulation of mitochondrial iron accumulation by Yfh1p, a putative homolog of frataxin. Science. 1997 Jun 13;276(5319):1709-12. doi: 10.1126/science.276.5319.1709. PMID 9180083
- [Background] Beal MF. Energetics in the pathogenesis of neurodegenerative diseases. Trends Neurosci. 2000 Jul;23(7):298-304. doi: 10.1016/s0166-2236(00)01584-8. PMID 10856939
- [Derived] Di Prospero NA, Sumner CJ, Penzak SR, Ravina B, Fischbeck KH, Taylor JP. Safety, tolerability, and pharmacokinetics of high-dose idebenone in patients with Friedreich ataxia. Arch Neurol. 2007 Jun;64(6):803-8. doi: 10.1001/archneur.64.6.803. PMID 17562928